CLINICAL TRIAL: NCT05834725
Title: A Pilot Randomized Controlled Trial of Resilience Coaching for Adolescents With Chronic Musculoskeletal Pain
Brief Title: Resilience Coaching for Adolescents With Chronic Musculoskeletal Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-020664; K23AR081409 (NIH)
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Pain, Chronic; Pain Syndrome; Psychological
Keywords: resilience coaching; chronic musculoskeletal pain
MeSH Terms: conditions — Chronic Pain; Somatoform Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resilience Coaching plus Usual Care (Experimental): Promoting Resilience in Stress Management (PRISM) is a 1:1, remotely delivered, resilience coaching program for adolescents with chronic illness, consisting of skill-building sessions in stress management, goal setting, cognitive re-framing, and benefit-finding. Sessions are held every 1-2 weeks for a total of 4 required and one optional session and each session lasts about 30-45 minutes.
  Interventions: Behavioral: Promoting Resilience in Stress Management
- Usual Care (Active Comparator): Usual care consists of an individualized treatment combining physical therapy, occupational therapy and psychological counseling. This is determined by the treating provider.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Promoting Resilience in Stress Management — Resilience coaching program.
  Arms: Resilience Coaching plus Usual Care
Other: Usual Care — Combination of physical therapy, occupational therapy, and psychological counseling as recommended by the treating provider.
  Arms: Usual Care

SUMMARY:
The goal of this clinical trial is to learn about resilience coaching in adolescents with chronic musculoskeletal pain. The main questions it aims to answer are to 1) determine how helpful resilience coaching is for teens with chronic musculoskeletal pain, 2) which participants are best suited for resilience coaching, and 3) barriers and facilitators to implementing resilience coaching as part of routine clinical care. Participants will complete survey measures and participate in the resilience coaching intervention called Promoting Resilience in Stress Management (PRISM). Researchers will compare youth in PRISM to those receiving usual care to determine whether PRISM leads to greater improvements in functional disability, psychological distress, and pain intensity than usual care alone.

DETAILED DESCRIPTION:
The purpose of this study is to find out if a resilience coaching program called Promoting Resilience in Stress Management (PRISM) can help youth with chronic musculoskeletal pain better cope with their chronic illness.Researchers will recruit a total of 130 youth with chronic musculoskeletal pain and one of their caregivers (total number of participants = 260). Teens will be randomly assigned to either a control group (usual care) or a treatment group (PRISM + usual care). PRISM consists of 4 study visits with a resilience coach, and one optional coming together session in which caregivers are invited to join. PRISM will occur over approximately 12 weeks. All participants will complete survey measures at baseline, 3-months and 9 months. Selected participants in PRISM will be invited to participate in interviews to provide feedback on the intervention. We will also interview 10 pediatric rheumatologists at other centers to obtain their feedback on the intervention and whether it would be valuable and feasible in their clinical setting. At the end of the study, researchers will assess whether participants in PRISM had improved functional disability, psychological distress and pain intensity as compared to the usual care arm.

ELIGIBILITY:
Inclusion Criteria:

* patient participants aged 12-17 years,
* newly diagnosed with chronic musculoskeletal pain, defined as bone, joint, muscle, or related soft tissue pain lasting ≥ 3 months
* willing to provide informed consent/assent
* one caregiver willing to consent and participate in dyad
* dyad identifies English as primary language
* mild or greater impairment due to pain (defined as Patient Reported Outcomes Measurement Information System Pain Interference T-score ≥ 60 at time of last clinic visit and/or self- or parent- reported impairment of activities of daily living due to pain at time of screening)

Exclusion Criteria:

* unable to provide assent and/or without a legal guardian able to provide consent for the study subject or themselves
* isolated/localized head pain or abdominal pain
* complex regional pain syndrome (CRPS)
* Receiving cognitive behavioral therapy at time of screening

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2025-11-02 (Actual); Study Completion 2026-06-14 (Estimated)

PRIMARY OUTCOMES:
Functional Disability | Measured at 3 months post-randomization.
  Functional disability at 3 months will be measured via the Functional Disability Inventory (FDI) score (ranging from 0-60 with higher scores indicating greater self-perceived functional disability).

SECONDARY OUTCOMES:
Psychological distress | Measured at 3 months post-randomization.
  Psychological distress at 3 months will be measured via the Kessler Psychological Distress Scale (K6) score. Responses are scored on 5-point Likert scale (total score ranging from 0-24). Previous studies have shown that scores ≥ 7 are consistent with "high" distress and those ≥ 13 meet criteria for serious, or debilitating psychological distress.
Pain intensity | Measured at 3 months post-randomization.
  Pain intensity at 3 months will be measured via the PROMIS (Patient Reported Outcome Measure Information System) Pediatric Numeric Rating Scale v1.0- Pain Intensity score (ranging from 0-10 with higher scores indicating greater pain intensity).

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Gmuca, MD MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gmuca S, Weiss PF, McGill M, Xiao R, Ward M, Nelson M, Sherry DD, Cronholm PF, Gerber JS, Palermo TM, Young JF, Rosenberg AR. The Feasibility and Acceptability of Resilience Coaching for Adolescent Chronic Musculoskeletal Pain: A Single-Arm Pilot Trial. Children (Basel). 2022 Sep 21;9(10):1432. doi: 10.3390/children9101432. PMID 36291374
- [Derived] Gmuca S, McGill M, Butler N, Xiao R, Cronholm PF, Young JF, Palermo TM, Weiss PF, Rosenberg AR. Resilience Coaching for Adolescent Chronic Musculoskeletal Pain: Protocol for a Pilot Randomized Controlled Trial of Promoting Resilience in Stress Management (PRISM). JMIR Res Protoc. 2025 Jul 22;14:e73385. doi: 10.2196/73385. PMID 40694836